CLINICAL TRIAL: NCT00237549
Title: The ADDITION Study. Anglo-Danish-Dutch Study of Intensive Treatment In PeOple With screeN Detected Diabetes in Primary Care
Brief Title: The ADDITION Study. Intensive Treatment in People With Screen Detected Diabetes in Primary Care.
Acronym: ADDTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Steno Diabetes Centre, Gentofte, Denmark (Unknown); University of Cambridge (Other); University Hospitals, Leicester (Other); Utrecht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: The ADDITION-study
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Screening; Intensive treatment; Polypharmacy; Primary care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): The 334 general practices in Denmark, United Kingdom and the Netherlands have been randomised to screening for diabetes followed by routine care (RC group) according to national guidelines, or screening followed by multifactorial treatment (IT group).
  Interventions: Procedure: optimised treatment

INTERVENTIONS:
Procedure: optimised treatment — The intervention targeted individual patients and the Primary Care Team. Practitioners were trained in a target driven, intensive multifactorial approach including lifestyle advice (smoking cessation, physical activity 30 min./day and healthy diet) and pharmacological treatment with the aim of reducing the complications of diabetes as described in protocol.
  The training included meetings, practice visiting, written feed back reports and reminders on controls.

SUMMARY:
The ADDITION study comprise 2 parts: screening for Type 2 diabetes and intensive treatment compared to standard treatment.

1. In the screening study, the feasibility and results of country specific models to identify undiagnosed individuals with Type 2 diabetes will be evaluated.
2. In the treatment study the effects of routine care in general practice according to local and national guidelines will be compared with an intensive ADDITION protocol, including structured lifestyle education (dietary modification, increased physical activity and smoking cessation) and intensive treatment of blood glucose, blood pressure and lipids, and prophylactic aspirin with or without motivational interviewing, on mortality, macrovascular and microvascular disease. Furthermore the impact of treatment on health status, treatment satisfaction and health service costs will also be assessed.

DETAILED DESCRIPTION:
Aims:

* To develop and evaluate strategies for early detection of type 2 diabetes in different countries and different populations.
* To study whether a multifactorial treatment strategy can reduce CVD-mortality and reduce the incidence of macro- and microvascular complications. The treatment strategy consists of motivational interviewing, encouraging behavioural changes (dietary advises, physical activity, smoking cessation) and intensive pharmacological treatment of blood pressure, blood glucose, and serum lipids
* To identify genetic markers predicting development of diabetic complications
* To evaluate health economical consequences of screening and early intervention for type 2 diabetes

Design and methods:

The study is an investigator initiated and designed study, initiated in Denmark by the two principal investigators, planned and conducted in collaboration between the four centers in Denmark, UK and the Netherlands. The study has two elements: a screening study and a subsequent intervention study.

In the screening study, the feasibility and results of country specific models to identify undiagnosed individuals with Type 2 diabetes will be evaluated.

In the treatment study the effects of routine care in general practice according to local and national guidelines will be compared with an intensive ADDITION protocol, including structured lifestyle education (dietary modification, increased physical activity and smoking cessation) and intensive treatment of blood glucose, blood pressure and lipids, and prophylactic aspirin with or without motivational interviewing, on mortality, macrovascular and microvascular disease. Furthermore the impact of treatment on health status, treatment satisfaction and health service costs will also be assessed.

Methodology - Screening study:

In Denmark > 300 primary care physicians from 5 different counties (Copenhagen, Aarhus, Ringkøbing, Ribe and Sønderjylland) participate in the study. Diabetes-related information is sent to all individuals aged 40-69 years enrolled in their practice. A questionnaire (diabetes risk score29) including age, gender, family history of type 2 diabetes; obesity; physical activity and previously diagnosed hypertension was used. Individuals scoring high on the questionnaire are encouraged to contact their physician for an examination of random blood glucose (RGB) and HbA1c. A step-wise strategy based on RBG, HbA1c, FPG and OGTT is used to diagnose diabetes In the Netherlands all people aged 50-69 years and listed with the participating primary care physicians is invited to fill in a diabetes risk questionnaire based on the same risk factors as in Denmark. Those at high risk of having type 2 diabetes are requested to come for a screening visit at a centre set up near the general practice. A stepwise screening strategy based on RBG, FPG and OGTT is used to diagnose diabetes In UK, different strategies are used in Cambridgeshire and Leicester. In Cambridgeshire a search of computerised general practice records is performed, using a simple validated risk score, based on routine general practice data (age, gender, prescribed medication and body mass index), to identify people in the age of 40-69 years at high risk of having undiagnosed diabetes30. Those with a high score undergo a stepwise screening strategy based on RBG, FPG and OGTT is used to diagnose diabetes In Leicester all white European subjects aged 40-75 years and Asian, black or Chinese subjects aged 25-75 years are invited in a restricted geographical region within Leicester. All attendant undergo an OGTT as the first screening step (unless FPG > 7.0 mmol/l)

Diagnostic procedures:

The diagnostic procedure includes a stepwise procedure minimizing the work-load on the general practitioner and includes the questionnaire, random capillary blood glucose and HbA1c as screening instruments followed by fasting capillary blood glucose (FCBG) and an oral glucose tolerance test in everyone with marginally elevated FCBG. The diagnostic criteria follow the most recent World Health Organization guidelines (31) and are based on two diagnostic glucose values measured on independent days.

Exclusion criteria:

Participants are excluded if they already have diabetes, are pregnant or lactating or have a severe psychotic illness, are house bound or have an illness with a likely survival of less than one year.

Outcome measures:

Outcome measures from the screening study include measures of the efficacy of the screening campaign, the objective health status of patients newly identified by the campaign, feasibility as reported by the primary care physician, and the economic impact or benefit of the a programme. Furthermore a substudy explores the psycho-social and ethical aspects of the screening programme.

Methodology - Intervention study:

All patients diagnosed as part of the screening programme are invited to enter the ADDITION-study. The study will include a minimum of 3000 patients with screen detected diabetes. The general practices are randomised to the routine care group (standard care as given by the GP) or to the intervention group which features a target driven, intensive multifactorial approach to treatment. The study is an open, multicentre, parallel group trial with randomisation of general practices. Patients are screened and recruited during the period January 1st 2000 and June 30th 2006. The end of follow up is by July 1st 2009. Participation is based on informed consent in accordance with the Declaration of Helsinki.

Intensive Treatment strategy:

The intensive multifactorial treatment includes lifestyle advices (concerning diet, physical activity, medication adherence and tobacco cessation), prescription of aspirin and stepwise increases in pharmacological treatment of blood glucose, blood pressure and lipids, according to strict targets (appendix 1). The treatment targets are as follows:

* HbA1c < 7.0
* Total cholesterol < 5.0 mmol/l (4.5 mmol/l if CVD present)but statin to everyone with total cholesterol > 3.5 mmol/l
* Blood pressure < 135/85
* Aspirin 75- 150 mg/day to everyone on antihypertensive treatment Behavioural advices include
* Smoking cessation
* Physical activity 30 min./day
* Healthy diet (low fat, 600g of fruit and vegetables/day)

The treatment targets may be intensified during the study according to the results of other clinical trials published during the study period, as the aim is to strive for treatment targets based on the most intensive guidelines available.

Within the intensive group a further randomisation allocates 50% of the patients to country specific interventions concerned with improving adherence to lifestyle changes and medication. This intervention, including the use of motivational interviewing) is delivered either by a trained facilitator (UK and The Netherlands) or through training of practitioners (Denmark), and is based on a client-centred non-directive counseling style to help patients explore and resolve ambivalence and stimulate lifestyle changes, appropriate diabetes self-care and adherence to medical treatment 32,33.

Pharmacological treatment:

The decision on which pharmaceutical drug to use for the individual patients with is made by the clinician as the study is target driven and not a trial comparing different specific drugs. The clinician is provided with recommendations for a treatment strategy (appendix 1), which should be based on balancing treatment effect, side-effects and cost. The main priority is achievement of treatment targets with a flexible lifestyle and low rates of side effects such as hypoglycaemia and weight gain.

Therapies are adjusted at 2 to 4-weekly intervals until targets are reached, thereafter every 3 months. HbA1c is taken every third month, in between antidiabetic drugs are adjusted according to blood glucose measurements in the interim.

Outcome measures: see other section.

Sample size and statistical power:

Based on levels of risk in the conservative-treatment arm of the UKPDS, the expected event rate is 3% per year for the combined endpoint (all-cause mortality, nonfatal myocardial infarction, stroke, revascularisation or amputation). With a sample size of 1350 patients in each arm (standard versus intensive treatment) the study will allow the detection of a 30% risk reduction in the intervention group at a significance level of 5% with a mean duration of follow-up of 5 years.

Timescale:

The screening study began in late 2000 and will end by June 30th 2006. Patients are enrolled into the treatment study following diagnosis in the screening study: thus the treatment study proceeds along with the evaluation phase of the screening study. The follow-up will continue until July 1st 2009.

Ethics and safety:

The Scientific Ethics Committee in the involved counties in Denmark and the Multipractice Study Committee have accepted the project, and the study has been approved by the ethical committees in UK and the Netherlands.

A data safety and monitoring committee will have access to all end point data (unblinded) after 1, 3 and 5 years, and the study will be terminated if the composite end point (including: Cardiovascular death, non-fatal MI, non-fatal stroke, revascularisation and amputation) should demonstrate a clear advantage of intensive versus standard treatment (p<0.001) or a clear advantage of the standard versus intensive treatment (p<0.01).

Perspectives of the trial:

The results of the study will be of immediate national and international relevance to policy decisions about screening for diabetes, and subsequent intensive treatment. If the study shows that screening and early intervention markedly reduces the risk of developing premature CVD, then the study will have potential important impact at the individual patient level as well as on the societal level. If the study fails to show an effect of screening and early intensive treatment then this would have direct impact on future recommendations for screening and treatment regimens, and the study could lead to significant savings if it shows that strict treatment targets are not essential in the early phase of the disease. The results of the sub-study will inform approaches to health promotion to the management of chronic disease and risk, and to strategies to support adherence applicable not only to diabetes but also to other chronic diseases.

References and Appendix 1 on www.addition.au.dk

ELIGIBILITY:
Inclusion Criteria:

Screening study: Every one aged 40-69 years (UK and DK) or 50-69 years(NL). Treatment study: All with screen detected type 2 diabetes.

Exclusion Criteria:

Participants are excluded if they already have diabetes at time of screening, are pregnant or lactating or have a severe psychotic illness, are house bound or have an illness with a likely survival of less than one year.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3057 (Actual)
Dates: Start 2001-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality | Sept 2010
MI (non fatal) | Sept 2010
Stroke (non fatal) | Sept 2010
Revascularisation (operating procedures) | Sept 2010
Amputations, non traumatic | Sept 2010

SECONDARY OUTCOMES:
All cause mortality | 2010
Development of renal impairment | 2010
Progression of retinopathy | 2010
Health economy, patient and health service costs and gains | 2010
Perceived health, SF36, AddQol | 2010
Neuropathy, periphery and autonomy | 2011

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Lauritzen, Professor, Study Chair — Institutute of Public Health, Dep. of General practice, Aarhus University, Denmark
Locations (4):
- Institute of Public Health, Aarhus, Aarhus, Denmark
- Julius Centre for health Sciences and Primary Care, University of Utrecht, Utrecht, Netherlands
- United Kingdom (2):
  - Department of Public Health and general Practice, Cambridge, Cambridge
  - University Hospital and Department of Health Sciences, University of Leicster, Leicester

REFERENCES:
- [Result] Lauritzen T, Griffin S, Borch-Johnsen K, Wareham NJ, Wolffenbuttel BH, Rutten G; Anglo-Danish-Dutch Study of Intensive Treatment in People with Screen Detected Diabetes in Primary Care. The ADDITION study: proposed trial of the cost-effectiveness of an intensive multifactorial intervention on morbidity and mortality among people with Type 2 diabetes detected by screening. Int J Obes Relat Metab Disord. 2000 Sep;24 Suppl 3:S6-11. doi: 10.1038/sj.ijo.0801420. PMID 11063279
- [Result] Sandbaek A, Griffin SJ, Rutten G, Davies M, Stolk R, Khunti K, Borch-Johnsen K, Wareham NJ, Lauritzen T. Stepwise screening for diabetes identifies people with high but modifiable coronary heart disease risk. The ADDITION study. Diabetologia. 2008 Jul;51(7):1127-34. doi: 10.1007/s00125-008-1013-0. Epub 2008 Apr 29. PMID 18443762
- [Result] Griffin SJ, Borch-Johnsen K, Davies MJ, Khunti K, Rutten GE, Sandbaek A, Sharp SJ, Simmons RK, van den Donk M, Wareham NJ, Lauritzen T. Effect of early intensive multifactorial therapy on 5-year cardiovascular outcomes in individuals with type 2 diabetes detected by screening (ADDITION-Europe): a cluster-randomised trial. Lancet. 2011 Jul 9;378(9786):156-67. doi: 10.1016/S0140-6736(11)60698-3. Epub 2011 Jun 24. PMID 21705063
- [Derived] Do DV, Han G, Abariga SA, Sleilati G, Vedula SS, Hawkins BS. Blood pressure control for diabetic retinopathy. Cochrane Database Syst Rev. 2023 Mar 28;3(3):CD006127. doi: 10.1002/14651858.CD006127.pub3. PMID 36975019
- [Derived] Bjerg L, Laugesen E, Andersen ST, Rosborg JF, Charles M, Vistisen D, Witte DR. Long-term effects of intensive multifactorial treatment on aortic stiffness and central hemodynamics after 13 years with screen-detected type 2 diabetes: the ADDITION-Denmark trial. Diabetol Metab Syndr. 2022 Aug 17;14(1):116. doi: 10.1186/s13098-022-00890-1. PMID 35978373
- [Derived] Griffin SJ, Rutten GEHM, Khunti K, Witte DR, Lauritzen T, Sharp SJ, Dalsgaard EM, Davies MJ, Irving GJ, Vos RC, Webb DR, Wareham NJ, Sandbaek A. Long-term effects of intensive multifactorial therapy in individuals with screen-detected type 2 diabetes in primary care: 10-year follow-up of the ADDITION-Europe cluster-randomised trial. Lancet Diabetes Endocrinol. 2019 Dec;7(12):925-937. doi: 10.1016/S2213-8587(19)30349-3. PMID 31748169
- [Derived] Lundgren JR, Faerch K, Witte DR, Jonsson AE, Pedersen O, Hansen T, Lauritzen T, Holst JJ, Vistisen D, Jorgensen ME, Torekov SS, Johansen NB. Greater glucagon-like peptide-1 responses to oral glucose are associated with lower central and peripheral blood pressures. Cardiovasc Diabetol. 2019 Oct 5;18(1):130. doi: 10.1186/s12933-019-0937-7. PMID 31586493
- [Derived] Simmons RK, Bruun NH, Witte DR, Borch-Johnsen K, Jorgensen ME, Sandbaek A, Lauritzen T. Does training of general practitioners for intensive treatment of people with screen-detected diabetes have a spillover effect on mortality and cardiovascular morbidity in 'at risk' individuals with normoglycaemia? Results from the ADDITION-Denmark cluster-randomised controlled trial. Diabetologia. 2017 Jun;60(6):1016-1021. doi: 10.1007/s00125-017-4230-6. Epub 2017 Mar 9. PMID 28280901
- [Derived] Charles M, Skriver MV, Griffin SJ, Simmons RK, Witte DR, Dalsgaard EM, Lauritzen T, Sandbaek A. Does Training and Support of General Practitioners in Intensive Treatment of People with Screen-Detected Diabetes Improve Medication, Morbidity and Mortality in People with Clinically-Diagnosed Diabetes? Investigation of a Spill-Over Effect in a Cluster RCT. PLoS One. 2017 Feb 2;12(2):e0170697. doi: 10.1371/journal.pone.0170697. eCollection 2017. PMID 28151941
- [Derived] Simmons RK, Borch-Johnsen K, Lauritzen T, Rutten GE, Sandbaek A, van den Donk M, Black JA, Tao L, Wilson EC, Davies MJ, Khunti K, Sharp SJ, Wareham NJ, Griffin SJ. A randomised trial of the effect and cost-effectiveness of early intensive multifactorial therapy on 5-year cardiovascular outcomes in individuals with screen-detected type 2 diabetes: the Anglo-Danish-Dutch Study of Intensive Treatment in People with Screen-Detected Diabetes in Primary Care (ADDITION-Europe) study. Health Technol Assess. 2016 Aug;20(64):1-86. doi: 10.3310/hta20640. PMID 27583404
- [Derived] den Ouden H, Berends J, Stellato RK, Beulens JW, Rutten GE. Effect of six years intensified multifactorial treatment on levels of hs-CRP and adiponectin in patients with screen detected type 2 diabetes: the ADDITION-Netherlands randomized trial. Diabetes Metab Res Rev. 2015 Oct;31(7):758-66. doi: 10.1002/dmrr.2669. Epub 2015 Jul 30. PMID 26109470
- [Derived] Kuznetsov L, Simmons RK, Sandbaek A, Maindal HT. The impact of intensive multifactorial treatment on perceptions of chronic care among individuals with screen-detected diabetes: results from the ADDITION-Denmark trial. Int J Clin Pract. 2015 Apr;69(4):466-73. doi: 10.1111/ijcp.12570. Epub 2014 Nov 7. PMID 25382351
- [Derived] Simmons RK, Carlsen AH, Griffin SJ, Charles M, Christiansen JS, Borch-Johnsen K, Sandbaek A, Lauritzen T. Variation in prescribing of lipid-lowering medication in primary care is associated with incidence of cardiovascular disease and all-cause mortality in people with screen-detected diabetes: findings from the ADDITION-Denmark trial. Diabet Med. 2014 Dec;31(12):1577-85. doi: 10.1111/dme.12574. Epub 2014 Sep 29. PMID 25185778
- [Derived] Dalsgaard EM, Vestergaard M, Skriver MV, Borch-Johnsen K, Lauritzen T, Sandbaek A. Socioeconomic position and cardiovascular risk factors among people with screen-detected Type 2 DM: six-year follow-up of the ADDITION-Denmark trial. Prim Care Diabetes. 2014 Dec;8(4):322-9. doi: 10.1016/j.pcd.2014.01.006. Epub 2014 Mar 6. PMID 24613817
- [Derived] Van den Donk M, Griffin SJ, Stellato RK, Simmons RK, Sandbaek A, Lauritzen T, Khunti K, Davies MJ, Borch-Johnsen K, Wareham NJ, Rutten GE. Effect of early intensive multifactorial therapy compared with routine care on self-reported health status, general well-being, diabetes-specific quality of life and treatment satisfaction in screen-detected type 2 diabetes mellitus patients (ADDITION-Europe): a cluster-randomised trial. Diabetologia. 2013 Aug 20;56(11):2367-77. doi: 10.1007/s00125-013-3011-0. Online ahead of print. PMID 23959571
- [Derived] Maindal HT, Toft U, Lauritzen T, Sandbaek A. Three-year effects on dietary quality of health education: a randomized controlled trial of people with screen-detected dysglycaemia (The ADDITION study, Denmark). Eur J Public Health. 2013 Jun;23(3):393-8. doi: 10.1093/eurpub/cks076. Epub 2012 Jun 13. PMID 23132875
- [Derived] Charles M, Fleischer J, Witte DR, Ejskjaer N, Borch-Johnsen K, Lauritzen T, Sandbaek A. Impact of early detection and treatment of diabetes on the 6-year prevalence of cardiac autonomic neuropathy in people with screen-detected diabetes: ADDITION-Denmark, a cluster-randomised study. Diabetologia. 2013 Jan;56(1):101-8. doi: 10.1007/s00125-012-2744-5. Epub 2012 Oct 12. PMID 23064291
- [Derived] Simmons RK, Sharp SJ, Sandbaek A, Borch-Johnsen K, Davies MJ, Khunti K, Lauritzen T, Rutten GE, van den Donk M, Wareham NJ, Griffin SJ. Does early intensive multifactorial treatment reduce total cardiovascular burden in individuals with screen-detected diabetes? Findings from the ADDITION-Europe cluster-randomized trial. Diabet Med. 2012 Nov;29(11):e409-16. doi: 10.1111/j.1464-5491.2012.03759.x. PMID 22823477
- [Derived] Johansen NB, Charles M, Vistisen D, Rasmussen SS, Wiinberg N, Borch-Johnsen K, Lauritzen T, Sandbaek A, Witte DR. Effect of intensive multifactorial treatment compared with routine care on aortic stiffness and central blood pressure among individuals with screen-detected type 2 diabetes: the ADDITION-Denmark study. Diabetes Care. 2012 Nov;35(11):2207-14. doi: 10.2337/dc12-0176. Epub 2012 Jul 11. PMID 22787176
- [Derived] Charles M, Ejskjaer N, Witte DR, Borch-Johnsen K, Lauritzen T, Sandbaek A. Prevalence of neuropathy and peripheral arterial disease and the impact of treatment in people with screen-detected type 2 diabetes: the ADDITION-Denmark study. Diabetes Care. 2011 Oct;34(10):2244-9. doi: 10.2337/dc11-0903. Epub 2011 Aug 4. PMID 21816977
- [Derived] Lauritzen T, Sandbaek A, Skriver MV, Borch-Johnsen K. HbA1c and cardiovascular risk score identify people who may benefit from preventive interventions: a 7 year follow-up of a high-risk screening programme for diabetes in primary care (ADDITION), Denmark. Diabetologia. 2011 Jun;54(6):1318-26. doi: 10.1007/s00125-011-2077-9. Epub 2011 Feb 22. PMID 21340624
- [Derived] Dalsgaard EM, Christensen JO, Skriver MV, Borch-Johnsen K, Lauritzen T, Sandbaek A. Comparison of different stepwise screening strategies for type 2 diabetes: Finding from Danish general practice, Addition-DK. Prim Care Diabetes. 2010 Dec;4(4):223-9. doi: 10.1016/j.pcd.2010.06.003. Epub 2010 Aug 1. PMID 20675208
- [Derived] Juul L, Sandbaek A, Foldspang A, Frydenberg M, Borch-Johnsen K, Lauritzen T. Adherence to guidelines in people with screen-detected type 2 diabetes, ADDITION, Denmark. Scand J Prim Health Care. 2009;27(4):223-31. doi: 10.3109/02813430903279117. PMID 19929182
- [Derived] Rubak S, Sandbaek A, Lauritzen T, Borch-Johnsen K, Christensen B. General practitioners trained in motivational interviewing can positively affect the attitude to behaviour change in people with type 2 diabetes. One year follow-up of an RCT, ADDITION Denmark. Scand J Prim Health Care. 2009;27(3):172-9. doi: 10.1080/02813430903072876. PMID 19565411
- See also: Study Website — http://www.addition.au.dk/